CLINICAL TRIAL: NCT01868074
Title: Enhancing Women's Health Through Assessing Foot Plasticity With Pregnancy
Brief Title: Study of Changes in the Feet With Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Neil A Segal, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201209787
Record Dates: First submitted 2013-05-23; First posted 2013-06-04 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Pregnancy
Keywords: pregnancy, arch height, collapsed arch
MeSH Terms: interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual (No Intervention): Participants who are not randomized to the fitted insole intervention
- Insole (Experimental): Participants randomized to use of a custom-molded insole during pregnancy
  Interventions: Device: Insole

INTERVENTIONS:
Device: Insole — Custom-molded arch-supporting insole
  Arms: Insole

SUMMARY:
This research is being conducted to determine whether use of an arch-supporting insole during pregnancy prevents alterations in foot structure and lower limb rotational movements. The investigators hypothesize that the arch collapse during pregnancy will be significantly reduced in women randomized to use the supportive insole compared with women randomized to the control group.

DETAILED DESCRIPTION:
Musculoskeletal impairments are a significant cause of functional limitations and disability in women. Women are at higher risk for osteoarthritis in comparison with men [1] and functional limitations due to arthritis are also more common in women. [2, 3] In addition, women are disproportionately affected (risk compared with men) by knee osteoarthritis (1.8x),[4] greater trochanteric pain syndrome (3.3x),[5] incident hip osteoarthritis[6] and chronic joint pain (1.3x),[7] including foot pain[8] knee pain[9] hip pain[9-12] and low back pain (1.2x).[7, 13] Preventing even a portion of these could avoid functional limitations and disability, enhance quality of life and result in considerable savings.[2] However, the etiology for the increased risk for these musculoskeletal diseases and impairments has not been elucidated.[1] Acute Changes in Foot Structure Are Reported with Pregnancy The disproportionate risk for these musculoskeletal problems may, in part, relate to biochemical and biomechanical changes that occur in a woman's body during pregnancy. For example, hallux valgus deformity, lateral deviation of the great toe often in conjunction with a bunion deformity, occurs in women at nine times the rate of men.[14] Both of these have been linked to reduction in arch height.[15] Body mass increases by an average of 9-13 kg during pregnancy.[16] There is also a seven to ten-fold increase in the relaxin level during pregnancy,[17-19] a peptide hormone produced by the corpus luteum which increases the flexibility and remodeling of collagen in central and peripheral joints in pregnant women.[17, 18, 20-26] Bearing increased weight on joints with increased laxity during pregnancy could potentially lead to permanent changes in the feet.[19, 26-28] Increases in foot length, width, and volume have been reported during pregnancy.[29, 30, 31] In addition to the anatomic changes in the foot, there are also changes in gait pattern during pregnancy.[32-35] Nyska found that the center of pressure on the foot during pregnancy shifts posteriorly to compensate for the increased anterior abdominal mass.[36] The combination of ligamentous laxity in the arch, increased body mass with pregnancy and the shift in the center of pressure towards the posterior part of the foot may potentially contribute to stretching of the ligaments supporting the arch, leading to loss of arch height.

More important than the foot changes that have been reported during pregnancy is the issue that these changes persist following completion of pregnancy. In a self-report study, we found a dose-response relationship between the number of pregnancies and the frequency of a report of a permanent change in foot size in women age 18-45.[37] We then conducted a longitudinal study to determine whether arch height loss both occurs and persists postpartum. Sixty women in their first trimester of pregnancy were enrolled and arch height and function were measured at baseline and approximately 19 weeks postpartum. There was a significant decrease in arch height and arch rigidity index at follow-up, with concomitant increases in foot length and arch drop. This study revealed that, not only was pregnancy associated with a permanent loss of arch height, but also the first pregnancy appeared to be the most significant with a reduction in arch rigidity (p<0.0001) and increases in foot length (p<0.0001), arch drop (p=0.0019) and center of pressure excursion during gait (p=0.0019). These changes in the feet could contribute to the increased risk for subsequent musculoskeletal disorders.

Arch Height Loss Leads to Adverse Biomechanical Changes at Other Joints Consideration of the effect of foot structure on forces and torques at other joints in the lower limb and spine as well as the need for energy generation and absorption by associated soft-tissue structures illustrates the importance of these potential changes. With each step, a series of events occurs that elicits biomechanical effects and compensations throughout the lower limb kinetic chain, in which movement at each joint influences movement at other joints in the chain.[38] Disruption of the complex interactions between skeletal, musculotendinous and ligamentous structures through loss of arch height may predispose to painful musculoskeletal conditions.[39-43] As the initial link in body loading during stance and movement, the feet are "where the rubber hits the road." The arch dynamically deforms to distribute the force, thereby absorbing the rapid impulse of loading. Changes in foot biomechanics that occur with changes in the foot structure alter the normal control of forces propagating from the foot to more proximal lower limb joints and the spine,[44] and contribute to pain in the feet, knees, hips,[41-43] and low back.

Possibly the most common cause of such changes in biomechanics is the loss of arch height. Excessive pronation strains the supporting structures of the foot and tendons that cross the ankle, leads to impaired balance,[45] can strain passive stabilizers such as the Achilles tendon, iliotibial band,[46] and anterior cruciate ligament,[47] and can contribute to permanent impairments in the soft tissue structures in the lower limbs.[47, 48] Thus, excessive pronation has been implicated in numerous musculoskeletal complaints, through pathologically re-distributing the ground reaction force over the foot,[49] changing patellar tracking in the femoral trochlea,[50] changing the angle of pull of muscular stabilizers in the lower limbs, and inducing a functional leg length inequality that alters hip and spine loading.[1] Therefore, there is a need to address this gap in knowledge to inform preventive interventions if there are musculoskeletal sequellae.

Biomechanical Changes Contribute to Musculoskeletal Disease Risk As mentioned previously, the permanent loss of arch height that occurs in about 40% of women with pregnancy leads to excessive pronation of the foot. This foot posture causes increased rotation of the tibia[51] and is communicated across the knee. These torques, in turn, may increase compressive and shear stress on the medial tibiofemoral and lateral patellofemoral compartments of the knee. This is important in light of previous work demonstrating that elevated contact stress is predictive of development of incident symptomatic knee osteoarthritis,[52] and the relative risk for knee replacement surgery increases with the number of pregnancies carried.[53] Closing Knowledge Gaps May Attenuate Musculoskeletal Disease Risk in Women In consideration of the evidence to date that pregnancy leads to a drop in the arch and that loss of the arch may contribute to musculoskeletal disease and disablement, there is a compelling rationale to characterize whether use of arch supports during pregnancy can prevent these adverse changes in foot structure during pregnancy. The proposed study will randomize women to either an arch-supportive insole or a control group(that does not wear insoles) and will measure static and dynamic arch structure in the early part of the first trimester and then again 8 weeks postpartum. Successful completion will inform the extent to which loss of arch height with pregnancy can be ameliorated using a conservative physical medicine intervention. This line of research holds great potential to inform preventive interventions to reduce the disproportionate risk for musculoskeletal disease and disability borne by women.

ELIGIBILITY:
Inclusion Criteria:

* Women in their first trimester of pregnancy
* Ages 18 and 40

Exclusion Criteria:

* lower limb joint or spinal surgery
* inflammatory joint or muscle problems such as rheumatoid or psoriatic arthritis
* diabetes
* collagen disorder such as Marfan Syndrome, Ehlers-Danlos Syndrome, Mixed Connective Tissue Disease, or Osteogenesis Imperfecta
* cannot walk without any assistance
* surgeries or have another medical condition that may affect their walking ability
* flat feet (absence of a longitudinal arch)
* inability to return for the follow-up visit 2 months after delivery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from clinics affliated with the University of Iowa Hospitals and Clinics; from the clniical trials Website; and from local day care facilities, schools, and pregnancy excercise classes.
  Exclusion criteria included women participating in in vitro fertilization, previous lower limb or spinal surgery, & chronic diseases.
Groups:
- Customized Insole Group: Each participant in the intervention group had her insole customized to fit her typical daily footwear and was instructed to wear the insoles as often as possible. Participants in the intervention group had their feet molded by a certified orthotist, using a 3M, soft cast. The casting was done in a non-weight bearing, hind-foot neutral position so the insoles would preserve the long transverse arch and maintain a biomechanically efficient state to control motion at the foot and ankle. These castings were used to custom form insoles with the following characteristics: Footlights athletic or dress model (per participant shoe preference), with 3/16" semi-rigid shells, no arch fill, extrinsic rearfoot and standard intrinsic forefoot posting. A research team member not involved with outcome measurements met with the participants to give them their insoles and confirm they fit.
- Usual Care Group: Participants in the control group were instructed to wear their usual footwear over the course of their pregnancy.
Period: Overall Study
Arm/Group | Customized Insole Group | Usual Care Group
Started | 36 | 36
Completed | 29 | 32
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Customized Insole: These participants were casted for customized insoles.
- Usual Care: Participants were instructed to wear their usual footwear over the course of their pregnancy.
- Total: Total of all reporting groups
Arm/Group | Customized Insole | Usual Care | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 30.2 (4.6) | 30.4 (4.4) | 30.3 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72
Foot Length Sitting [Mean (Standard Deviation); unit: mm] | 240.4 (13.5) | 240.1 (10.2) | 240.25 (11.85)
Foot Length Standing [Mean (Standard Deviation); unit: mm] | 242.8 (10.2) | 243.0 (13.7) | 242.9 (11.95)
AHI Sitting [Mean (Standard Deviation); unit: ratio] — The arch height index (AHI) was calculated as the dorsum height at 50% of total foot length divided by the ipsilateral truncated foot length.
  ratio | 0.35 (0.02) | 0.35 (0.02) | 0.35 (0.02)
AHI Standing [Mean (Standard Deviation); unit: ratio] — The arch height index (AHI) was calculated as the dorsum height at 50% of total foot length divided by the ipsilateral truncated foot length.
  ratio | 0.33 (0.02) | 0.33 (0.02) | 0.33 (0.02)
Arch Drop [Mean (Standard Deviation); unit: mm] — Arch drop was calculated by subtracting the standing arch height from the seated arch height.
  mm | 3.0 (1.4) | 2.8 (1.1) | 2.9 (1.3)
Arch Rigidity [Mean (Standard Deviation); unit: ratio] — The arch rigidity index, a measure of the ability of the foot to maintain the arch when weight-bearing, was determined by dividing the standing AHI by the seated AHI. A value of 1.0 would indicate a perfectly rigid arch, while smaller values would indicate a more flexible arch.
  ratio | 0.94 (0.03) | 0.94 (.02) | 0.94 (0.03)
Center of Pressure Excursion Index at self-selected speed [Mean (Standard Deviation); unit: ratio] — The Center of Pressure Excursion Index is a measurement of the lateral displacement of the center of pressure curve from a reference line drawn from the initial to the final centers of pressure during stance phase of gait, and standardized to the width of the anterior third of the foot during pedobarography.
  ratio | 18.6 (6.2) | 21.3 (6.3) | 19.95 (6.25)
Center of Pressure Excursion Index (3mph) [Mean (Standard Deviation); unit: ratio] | 18.1 (5.9) | 20.8 (6.6) | 19.9 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Arch Drop
Description: Measurement of Arch Drop (Sitting arch height minus standing arch height) using Arch Height Index Measurement System
Time Frame: baseline, 8 weeks postpartum
Measure: Mean (Standard Error); unit: mm
Groups:
- Customized Insole Group: This intervention group were casted for customized insoles.
- Usual Care Group: Participants in the control/usual group were instructed to wear their usual footwear over the course of their pregnancy.
Arm/Group | Customized Insole Group | Usual Care Group
Number analyzed (Participants) | 29 | 32
mm | -.02 (.15) | .07 (.14)

2. Secondary Outcome: Change in Arch Rigidity
Description: The arch rigidity index, a measure of the ability of the foot to maintain the arch when weight-bearing, was determined by dividing the standing AHI by the seated AHI. A value of 1.0 would indicate a perfectly rigid arch, while smaller values would indicate a more flexible arch.
Time Frame: baseline, 8 weeks postpartum
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Customized Insole Group | Usual Care Group
Number analyzed (Participants) | 29 | 32
ratio | 0 (0) | 0 (0)

3. Secondary Outcome: Change in CPEI (3mph)
Description: The Center of Pressure Excursion Index (CPEI) is a measurement of the lateral displacement of the center of pressure curve from a reference line drawn from the initial to the final centers of pressure during stance phase of gait, and standardized to the width of the anterior third of the foot during pedobarography.
Time Frame: baseline, 8 weeks postpartum
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Customized Insole Group | Usual Care Group
Number analyzed (Participants) | 29 | 32
ratio | .21 (.56) | -.02 (.53)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored monthly.
Description: Participants completed a web questionnaire regarding comfort with the insoles, foot pain and knee pain.
Arm/Group | Customized Insole | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No